CLINICAL TRIAL: NCT00089323
Title: Bone Marrow Analysis In Early-Stage Breast Cancer
Brief Title: Diagnostic Procedures in Detecting Tumor Cells in the Bone Marrow of Patients Undergoing Surgery for Stage I, Stage II, or Stage IIIA Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NSABP BP-59; NSABP-BP-59
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage II breast cancer; stage IIIA breast cancer; male breast cancer; stage IB breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1: Bone Marrow Aspiration (Other)
  Interventions: Procedure: Bone Marrow Aspiration

INTERVENTIONS:
Procedure: Bone Marrow Aspiration

SUMMARY:
RATIONALE: Diagnostic procedures that detect tumor cells in the bone marrow may help doctors predict disease recurrence and plan more effective treatment.

PURPOSE: This clinical trial is studying how well diagnostic procedures work in detecting tumor cells in the bone marrow of patients who have undergone surgery for stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the relative risk of death associated with the presence of tumor cells in the bone marrow of patients with stage I, II, or IIIA breast cancer undergoing surgery and bone marrow analysis using multicolor fluorescence immunocytochemistry and bright field immunocytochemistry.

Secondary

* Compare multicolor fluorescence immunocytochemistry vs bright field immunocytochemistry in the detection of bone marrow micrometastases in these patients.

OUTLINE: This is a multicenter study.

Patients undergo bone marrow aspiration during surgical resection of the primary tumor. Bone marrow cells and tumor samples are analyzed using bright field immunocytochemistry and multicolor fluorescence immunocytochemistry.

Patients are followed every 12 months for up to 10 years.

PROJECTED ACCRUAL: A total of 1,634 patients will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion criteria

* Histologic diagnosis of invasive adenocarcinoma of the breast diagnosed by core, incisional, or excisional biopsy.
* All of the following staging criteria must be met: Primary tumor must be operable and staged as cT1-3 by clinical evaluation. Ipsilateral nodes must be cN0-1 by clinical evaluation. No evidence of metastatic disease (M0).

Exclusion criteria:

* Patients with any history of breast malignancy including DCIS (patients with a history of Lobular Carcinoma in Situ (LCIS) are eligible).
* Treatment including radiation therapy, chemotherapy, and/or hormonal therapy administered for the currently diagnosed breast cancer prior to study entry. The only exception is hormonal therapy, which may have been given for up to a total of 28 days after diagnosis and before study entry.
* Patients who will be receiving preoperative chemotherapy.
* Bilateral malignancy (including DCIS).
* Other non-breast malignancies unless the patient is considered disease-free for 5 years before study entry and is deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, melanoma in situ, colon carcinoma in situ, and basal cell and squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1630 (Actual)
Dates: Start 2007-01; Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | From time of randomization to death from any cause through 10 years.

SECONDARY OUTCOMES:
Tumor cell presence as measured by bright-field and multicolor fluorescence immunocytochemical methods | As detected at time of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (53):
- United States (49):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Morton Plant Hospital, Clearwater, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Union Hospital of Cecil County, Elkton, Maryland
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - United Hospital Center, Clarksburg, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (4):
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHUM - Hotel Dieu Hospital, Montreal, Quebec
  - CHUM - Hopital Saint-Luc, Montreal, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec